CLINICAL TRIAL: NCT02828501
Title: Additive Effects of Combined Cervical and Lumbar Manipulation on Pain Pressure Threshold in a Single Session
Brief Title: Additive Effects of Combined Spinal Manipulations on Pain Pressure Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Max Jordon, PhD Candidate, University of South Carolina
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00043661
Record Dates: First submitted 2016-06-22; First posted 2016-07-11 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Pain Threshold
Keywords: Pain Threshold
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lumbar manipulation group (Experimental): Spinal Manipulation
  Interventions: Procedure: Spinal Manipulation
- Cervical manipulation group (Experimental): Spinal Manipulation
  Interventions: Procedure: Spinal Manipulation
- Control group (No Intervention): This group will receive a 2 minute supine rest between measurements

INTERVENTIONS:
Procedure: Spinal Manipulation — A spinal manipulation is a high velocity, low amplitude thrust through a physiological barrier in order to elicit a cavitation.
  Arms: Cervical manipulation group; Lumbar manipulation group

SUMMARY:
Physical therapists frequently use spinal manipulation therapy (SMT) to treat spinal pain. However, the methods by which SMT exerts its effects are not well understood. The aim of this study is to assess potential changes in pain pressure threshold following both a cervical and lumbar spine manipulation in a single treatment session at sites local and diffuse to the site of manipulation application. This study will also attempt to determine if the order of the cervical and lumbar manipulation application impacts pain pressure threshold changes.

DETAILED DESCRIPTION:
The aim of the proposed study is to add to the literature pertaining to the effects of spinal manipulation on PPT. To date, no studies have assessed whether or not there is an additive effect of multiple manipulations during a single treatment session on PPT. The proposed study will assess potential changes in PPT between baseline measurements, following a single cervical or lumbar manipulation, and after the delivery of second spinal manipulation performed on a different segment. The study design will allow for the investigation of possible additive effects, as well as for the effect of the first manipulation to be assessed independently of the second. Order of delivery of the cervical and lumbar manipulation will be randomized among participants to allow investigators to consider the possibility that the order of the manipulations impacts PPT changes.

Research Questions

1. Is a single spinal manipulation of either the cervical or lumbar spine associated with an immediate increase in pain pressure threshold either locally or diffusely when compared to a no treatment control?
2. What is the effect of a second spinal manipulation at a different segment immediately following the first spinal manipulation on pain pressure threshold?
3. Is there a difference based on the order of which spinal manipulation is administered (cervical first, then lumbar; lumbar first, then cervical) on post-intervention local and diffuse pain pressure threshold?

Overview of Research Design This study will be a cross-sectional, single-blinded randomized control trial. This will be a single session, experimental approach in which participants who meet the inclusion/exclusion criteria will be divided into three groups: treatment group 1, treatment group 2, and control group. Group assignment will be performed using randomized concealed allocation. Participants will undergo pain pressure threshold testing using pressure algometry, followed by a cervical manipulation for treatment group 1 and a lumbar manipulation for treatment group 2. The control group will rest quietly for an allotted amount of time. Upon completion of the first intervention, a second pain pressure threshold assessment will be performed. Treatment group 1 will then receive a lumbar manipulation, while treatment group 2 receives a cervical manipulation. The control group will again rest quietly. Following the second intervention, a final pain pressure threshold assessment will be taken. The primary dependent measures will be 1) current pain intensity as reported by a verbal numeric pain rating scale, 2) self-reported stiffness, and 3) pain pressure threshold measured in Newtons.

ELIGIBILITY:
Inclusion Criteria:

* To be included in this study, consenting male and female participants must be between the ages of 18 and 60. This age range insures skeletal maturity with a reasonably low prevalence of severe osteoarthritis or osteopenia.

Exclusion Criteria:

* The presence of any of the following factors will exclude the participant from this study:

  1. Currently involved in a worker's compensation claim or in personal injury litigation.
  2. Currently on, or applying for, permanent or temporary disability due to a medical or mental health condition.
  3. Currently taking prescription analgesics.
  4. Activity-limiting pain arising from any site other than listed in the specific entry criteria.

Additional exclusion criteria include the presence of any of the following conditions as determined by prior medical and/or radiographic examination or initial MRI:

* pregnancy or have been pregnant in the last year;
* spinal osteoporosis or osteopenia;
* inflammatory joint disease;
* an infection involving the spine;
* severe arthritis;
* any current (within 5 years) neoplastic condition;
* any history of vertebral fracture with current bony instability or measurable deformity;
* severe lumbar stenosis (defined as an A-P diameter of the thecal sac of less than 5 mm at any level, from mid-sagittal lumbar T2-weighted MRI);
* diagnosis of cervical spinal stenosis
* any abnormalities or compression of the spinal cord, cauda equine, or spinal nerves;
* any upper or lower extremity nerve impairment;
* unstable angina, congestive heart failure, orthopnea, or severe hypertension;
* any history of a surgical procedure to the cervical or thoracic or lumbar spine;
* any surgical procedures to the abdomen, thorax, upper extremities, head or neck in the past 6 months prior to enrollment in the study;
* history of whiplash in the last 6 weeks;
* evidence of central nervous system involvement, to include hyperreflexia, sensory disturbances, unsteadiness during walking, nystagmus, loss of visual acuity, impaired sensation of the face, altered taste, the presence of pathological reflexes (i.e. positive Hoffman's and/or Babinski reflexes), etc.;
* resting blood pressure greater than 140/90 mmHg at initial intake;
* presence of any of the following atherosclerotic risk factors: hypertension, diabetes, heart disease, stroke, transient ischemic attack, peripheral vascular disease, smoking, hypercholesterolemia, or hyperlipidemia;
* current use of any of the following medications: narcotics, opiate-based analgesics, prescribed anticoagulants (this does not include low doses of ASA or NSAIDs), and oral or injected corticosteroids.

These criteria are designed to exclude individuals for whom spinal manipulation is contraindicated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2015-03; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Pressure-Pain Threshold as assessed by a pressure algometer | Two minutes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jordon MK, Beattie PF, D'Urso S, Scriven S. Spinal manipulation does not affect pressure pain thresholds in the absence of neuromodulators: a randomized controlled trial. J Man Manip Ther. 2017 Sep;25(4):172-181. doi: 10.1080/10669817.2016.1230352. Epub 2016 Sep 12. PMID 28912629